CLINICAL TRIAL: NCT05220748
Title: A Phase 1 First-in-Human, Drug-dose Escalation Study of RM-1995 Photoimmunotherapy, as Monotherapy or Combined With Pembrolizumab, in Patients With Advanced Cutaneous Squamous Cell Carcinoma or With Head and Neck Squamous Cell Carcinoma
Brief Title: RM-1995 Photoimmunotherapy, as Monotherapy or Combined With Pembrolizumab, in Patients With Advanced CuSCC and HNSCC
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Decision was made due to a strategic re-evaluation of pipelines; no patients were enrolled.
Sponsor: Rakuten Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RM-1995-101
Record Dates: First submitted 2022-01-11; First posted 2022-02-02 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Cutaneous Squamous Cell Carcinoma; Head and Neck Squamous Cell Carcinoma
Keywords: Rakuten Medical; RM-1995; RM-1995-101; HNSCC; CUSCC; head and neck squamous cell carcinoma; cutaneous squamous cell carcinoma; PIT; photoimmunotherapy; skin cancer; skin; head and neck cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Skin Neoplasms; Head and Neck Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- RM-1995 Photoimmunotherapy (Phase 1a Monotherapy) (Experimental): Patients with locally advanced cuSCC or HNSCC or metastatic disease that has recurred or progressed, despite all available standard therapies.
  Interventions: Combination Product: RM-1995
- RM-1995 Photoimmunotherapy + Pembrolizumab (Phased 1b Combination Therapy) (Experimental): Patients with locally advanced cuSCC or HNSCC or metastatic disease that has recurred or progressed, despite all available standard therapies.
  Interventions: Combination Product: RM-1995; Biological: Pembrolizumab

INTERVENTIONS:
Combination Product: RM-1995 — RM-1995 will be administered by intravenous (IV) infusion followed approximately 24 hours later by tumor illumination with 690 nm non thermal red light using the PIT690 Laser System. The starting dose of RM-1995 will be 0.25 mg/kg and escalated up to 2.0 mg/kg over 6 dosing cohorts
Biological: Pembrolizumab — Pembrolizumab (200 mg) will be administered by intravenous (IV) infusion one week before the first RM-1995 PIT treatment and the second dose three weeks later for patients in the combination arm. Once the DLT window is complete, pembrolizumab dosage will be maintained at either 200 mg Q3w, or shift to 400 mg Q6w, per investigator discretion.
  Arms: RM-1995 Photoimmunotherapy + Pembrolizumab (Phased 1b Combination Therapy)

SUMMARY:
A phase 1a/1b, open-label, RM-1995 drug-dose escalation study designed to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary efficacy of RM-1995 photoimmunotherapy treatment as monotherapy (phase 1a) or combined with pembrolizumab (phase 1b) in patients with cutaneous squamous cell carcinoma (cuSCC) or head and neck squamous cell carcinoma (HNSCC) that has progressed despite all available standard therapies.

DETAILED DESCRIPTION:
Enrollment consists of six cohorts of patients with locally advanced cuSCC or HNSCC that has recurred or progressed on or after at least one prior line of therapy, which must include prior platinum-based chemotherapy and is not eligible for further locoregional therapy, or with metastatic disease that has recurred or progressed after all available standard therapies. Patients will receive anti-CD25 antibody, conjugated to the light-activatable dye, IRDye® 700DX, followed by illumination with non-thermal red light (RM-1995 photoimmunotherapy)) as monotherapy (phase 1a), or in combination with pembrolizumab (phase 1b).

Patients are required to have measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1,Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2, and a superficial lesion accessible to photoimmunotherapy at the time of screening.

Phase 1a primary objectives are to evaluate the safety and tolerability of RM-1995 photoimmunotherapy treatment as monotherapy and determine the maximum tolerated dose (MTD) or maximum administered dose (MAD).

Phase 1b primary objectives are to evaluate the safety and tolerability of RM-1995 photoimmunotherapy treatment in combination with pembrolizumab and determine the MTD or MAD.

ELIGIBILITY:
* Inclusion Criteria. Patients must meet all the following criteria to be eligible to participate in the study:
* Patient must be at least 18 years old.
* Patient must have tumor types of head and neck squamous cell carcinoma (HNSCC), cutaneous squamous cell carcinoma (cuSCC)
* Locally advanced or locoregional disease that has recurred or progressed on or after at least one prior line of therapy, which must include prior platinum-based chemotherapy, and is not eligible for further locoregional treatment (ie, standard surgery or radiation), or for which locoregional treatment has proved to be intolerable or is medically contraindicated.
* Metastatic disease that has recurred or progressed following prior platinum-based chemotherapy, prior immunotherapy with PD-(L)1 inhibitors, or other standard of care systemic treatment, has proven to be ineffective, intolerable, or is considered medically contraindicated in the opinion of the Investigator
* Patient must have tumors with at least one superficial lesion of the skin or oral cavity, not deeper than 1 cm and that is accessible for photoimmunotherapy treatment. Note: Lesions that are in the pharynx and larynx will not be included in the treatment.
* Patient must have the ability to provide representative tumor specimens with an associated pathology report.
* Patient must have measurable disease by RECIST 1.1 as assessed by Investigator.
* Patient must have ECOG performance status of 0 to 2 at the time of screening
* Patient has life expectancy ≥ 3 months based on Investigator's judgement.
* Adequate organ function laboratory values (Hematology, Hepatic, Renal and Coagulation).
* Female patients of childbearing potential must not be pregnant or breastfeeding and must be willing to use 2 methods of highly effective birth control, or practice abstinence throughout the study and for at least 120 days after the last dose of study medication.
* Male patients must be sterile or agree to use an adequate method of contraception or practice abstinence starting with the first dose of study medication and for at least 120 days after the last dose of study medication.

Exclusion Criteria. Patients who meet any of the criteria below will be ineligible to participate in the study:

* Receiving any other investigational agents, approved anticancer therapies, including chemotherapy, hormonal therapy, ultraviolet-light therapy, or other topical therapy within 2 weeks or 5 half-lives, whichever is longer, before initiation of study treatment, with the following exceptions:
* Hormone-replacement therapy or oral contraceptives
* Herbal therapy, including herbal therapy intended as anticancer therapy and medicinal cannabinoids taken to reduce symptom burden, must be discontinued at least 1 week before the first dose of pembrolizumab (combination therapy) or the first dose of RM-1995 (monotherapy)
* Palliative radiotherapy for painful boney metastases or metastases in potentially sensitive locations (eg, epidural space) must be completed > 2 weeks before the first dose of pembrolizumab (combination therapy) or the first dose of RM 1995 (monotherapy)
* Previously initiated bisphosphonate or denosumab therapy for bone metastases may be continued during study participation.
* Treated with local radiation therapy within 12 weeks before the first dose of study treatment. Patients must have recovered from all radiation-related toxicities to Grade < 1 or baseline and must not require steroids.
* Treatment with systemic immunostimulatory agents not described above (including but not limited to IFN-α, IL-2) within 6 weeks or 5 half-lives of the drug, whichever is shorter, before the first dose of study treatment.
* Adverse events from prior anticancer therapy that have not resolved to Grade ≤ 1, except for alopecia or endocrinopathy managed with replacement therapy.
* Patients who have tumors at sites that may compromise sensitive and vital anatomic structures.
* Malignancies other than disease under study within 3 years prior to treatment start, except for those with a negligible risk of metastasis or death.
* Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within the previous 3 months, unstable arrhythmias, or unstable angina.
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis, cirrhosis, or inherited liver disease.
* Prior allogeneic bone marrow transplantation or prior solid organ transplantation.
* Known history of testing positive for human immunodeficiency virus or acquired immunodeficiency syndrome -related illness.
* Known infection or detection of active Hepatitis B (e.g., HBsAg positive), Hepatitis C (eg, RNA [qualitative]), or SARS-CoV-2 (qualitative).
* Received a live, attenuated vaccine within 4 weeks before the first dose of study treatment or anticipating the receipt of a required live, attenuated vaccine during the study (based on known medical history).
* Receiving drugs known to prolong the QTc interval while on study treatment or within 14 days before the first dose of study treatment.
* Receiving cytochrome P450 (CYP) substrates, inhibitors, inducers while on study treatment or within 14 days before the first dose of study treatment.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or poorly controlled psychiatric illness.
* Received oral or IV antibiotics within 2 weeks before the first dose of study treatment
* Major surgery or significant traumatic injury within 28 days before the first dose of study treatment or anticipation of the need for major surgery that is unrelated to study intervention during the study.
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to any of the components of RM-1995 or to other recombinant chimeric, human, or humanized antibodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Phase 1a Monotherapy: Evaluate the safety and tolerability of RM-1995 PIT treatment, and determine the Maximum Tolerated Dose (MTD) or Maximum Administered Dose (MAD). | 24 months
  Incidence of dose-limiting toxicities (DLTs), frequency of adverse events, and MTD or MAD
Phase 1b Combination Therapy: Evaluate the safety and tolerability of RM-1995 PIT treatment in combination with pembrolizumab and determine the MTD or MAD. | 24 months
  Incidence of dose-limiting toxicities (DLTs), frequency of adverse events, and MTD or MAD

SECONDARY OUTCOMES:
Serum concentration of RM-1995. | Various timepoints from Cycles 1, 2, and 3, Day 1 through Day 21. Each cycle is 21 days.
Serum concentration of total antibody. | Various timepoints from Cycles 1, 2, and 3, Day 1 through Day 21. Each cycle is 21 days.
Serum concentration of IR-700. | Various timepoints from Cycles 1, 2, and 3, Day 1 through Day 21. Each cycle is 21 days.
Assess antitumor activity of RM-1995. | 24 months
  Objective Response Rate (ORRPIT) defined as the proportion of patients with confirmed PIT-treated tumor response of complete response or partial response per RECIST 1.1 (or irRECIST for patients receiving pembrolizumab combination therapy)

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Schechter, Study Chair — Rakuten Medical, Inc.

IPD SHARING:
Plan to Share IPD: No